CLINICAL TRIAL: NCT00345150
Title: Phase 1 Study of the Effects of Systemic Nitric Oxide Inhibition With Ng-Monomethyl-L-Arginine on Renal Hemodynamics and Sodium Excretion in Patients With Essential Hypertension and Healthy Controls
Brief Title: Effects of Inhibition of NO-Synthesis on Renal Hemodynamics and Sodium Excretion in Patients With Essential Hypertension and Healthy Controls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: MED.RES.HOS.1995.01.JNB
Record Dates: First submitted 2006-06-24; First posted 2006-06-27 (Estimated); Last update posted 2006-06-27 (Estimated); Status verified 2006-06

CONDITIONS: Hypertension
Keywords: hypertension; nitric oxide; renal hemodynamics
MeSH Terms: conditions — Hypertension | interventions — omega-N-Methylarginine; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Ng-monomethyl-L-arginine (drug)

SUMMARY:
The study tests the hypothesis that systemic and renal nitric oxide synthesis is changed in essential hypertension by investigating the effects of a non selective nitric oxide inhibitor on renal hemodynamics and sodium excretion in patients with essential hypertension. The results are compared with a group of healthy subjects.

DETAILED DESCRIPTION:
The study investigates the effects of Ng-monomethyl-L-arginine (L-NMMA) on:

1. renal hemodynamics (renal plasma flow and glomerular filtration rate)
2. renal sodium excretion
3. lithium clearance and fractional lithium excretion
4. plasma levels of vasoactive hormones
5. blood pressure and heart rate

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension (blood pressure > 140/90) with no signs of secondary hypertension
* P-creatinine < 200 µmol/L

Exclusion Criteria:

* Anamnestic or clinical signs of heart disease, renal disease, liver disease, neoplastic disease, anemia or cerebro-vascular insult
* Medication except antihypertensives
* Drug or alcohol abuse
* Pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Overall Officials: Jesper N Bech, MD, Ph.D., Principal Investigator — Dept. of Medicine, Holstebro Hospital, 7500 Holstebro, Denmark; Erling B Pedersen, Professor, Study Chair — Holstebro Hospital, 7500 Holstebro, Denmark